CLINICAL TRIAL: NCT06639438
Title: Molecular and Behavioral Characterization of Post-Operative Sensory Outcomes in Individuals With Chronic Pain or Persistent Opioid Use
Brief Title: Sensory Outcomes in Active Substance Users
Status: Recruiting | Type: Observational
Sponsor: Boston Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: H-44193
Record Dates: First submitted 2024-10-07; First posted 2024-10-15 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Post Operative Pain; Opioid Use, Unspecified
Keywords: Opioid use disorder (OUD); Gene expression; Visium slide sequencing; Inflammatory profile; Sensation pain; Flow cytometry
MeSH Terms: conditions — Pain, Postoperative; Opioid-Related Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A 10 ml blood sample will be collected for serum analysis immediately before, during, and 24 hours after the surgical procedure. During the procedure, A 5mm (length) x 3mm (width) x 2 mm (depth) tissue sample from the incision site will be collected for later spatial transcriptomic analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group 1- Patients with Opioid Use Disorder (OUD): Participants in this group will be diagnosed with OUD, defined by cognitive, behavioral, and physiological symptoms indicating using opioids despite significant opioid-related problems.
- Group 2- Patients who are engaged in long-term opioid therapy (LTOT) for chronic pain: Participants in this group will be engaged in long-term opioid therapy (LTOT) for chronic pain management under medical supervision, without exhibiting the problematic behaviors or experiencing the significant impairment or distress outlined in the OUD criteria.
- Group 3- Patients with chronic pain but no (or minimal) opioid use: Participants in this group will have chronic pain but no (or minimal) opioid use where chronic pain is defined as pain that lasts more than three months or beyond the expected period of healing but opioid use is < 20MME with <3 weeks of duration.
- Group 4- Patients without chronic pain: Participants in this group will not suffer from chronic pain but choose to undergo spine surgery due to structural abnormalities or conditions that could potentially lead to pain, neurological issues, or other significant health problems

SUMMARY:
The incidence and severity of postoperative pain after spine surgery are notably high, often requiring intensive management and potentially affecting the patient's recovery, satisfaction, and long-term outcomes. Post-operative pain is particularly difficult to manage in patients with substance use disorder likely due to a combination of withdrawal symptoms and molecular changes in the pain matrix. Opiates are the leading cause of overdose related fatalities, and carry a significant burden of substance related morbidity and mortality. As over 80% of patients undergoing low-risk surgery receive opioid prescriptions, the investigators aim to identify unique molecular characteristics of pain within current and previous opioid users, which have been understudied in this context. This study also seeks to understand the molecular mechanisms underlying worsened postoperative pain in patients with opioid use disorder (OUD).

Flow cytometry analysis of human serum will be done, which will assess circulating immune cells that can contribute to exacerbated surgery site inflammation. Spatial profiling of gene expression will be done in the dermis using Visium slide sequencing, focusing on the interplay between nerve endings, resident immune cells, and supporting dermal cells, all of which collectively contribute to the sensation pain. Both the visual pain rating scale and McGill Pain Questionnaire will be used to comprehensively quantify pain outcomes during the participant's postoperative recovery stay after surgery in an effort to better understand postoperative pain management with biomarkers of worsened postoperative pain.

DETAILED DESCRIPTION:
The objective for this research are:

1. Assess differences in pain reception in patients with existing or previous opioid use disorder versus controls after elective spine surgery via pain questionnaires at multiple time points during the perioperative care.
2. Assess circulating immune signatures and neuropeptides associated with pain signaling before and after surgery in patients with and without OUD using flow cytometry and ELISA of patient serum.
3. Assess molecular signatures of dermal cells and nerve endings patients with and without OUD using spatial transcriptomics on epidermis- and dermis-containing tissue samples from surgical incision.

ELIGIBILITY:
Inclusion Criteria:

Opioid user cohorts:

* Individuals with current OUD as defined by The Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5)
* Individuals requiring ≥20 mg of MME/day medication to manage a chronic pain problem.
* Patients scheduled to undergo elective surgery
* Able to provide informed consent

Control Group Cohorts:

* Individuals who are not taking high dose opioids (≤20 MME/day) nor illicit substances and have no history of opioid use disorder
* Individuals with reported chronic pain not yet taking medication for their pain
* Patients scheduled to undergo elective surgery
* Able to provide informed consent

Exclusion Criteria:

Substance User Cohort:

* Patients with contraindications for elective surgery
* Individuals with no history of opioid use

Control Group Cohort:

* Individuals with a history of opioid use >20 MME/day or illicit substance use
* Patients with contraindications for elective surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with elective spine procedures scheduled involving incision (including laminectomy, discectomy, foraminotomy, scoliosis correction, decompression and fusion) will be divided into four groups: two no opiod use groups and two opioid use groups. The no opioid use groups will consist of two subgroups of participants with no prior pain disorders who have received no long-term opioid prescriptions (n=10), as well as patients with chronic pain disorders who have received no long-term high dose opioid prescriptions (n=10). The opioid use group will consist of two subgroups- participants with OUD (n=10), and participants without OUD, but have been prescribed opioid medication for chronic pain disorders (n=10).
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-02-02 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Specific gene expressed | The date of scheduled surgery assessed through the study completion, about two years
  This outcome will be assessed by the transcriptomic profile of dermal tissue from patient excision site using the Visium system to quantify gene expression changes in the dermis. Dermis tissue, about 5mm (length) x 3mm (width) x 2 mm (depth) in size, will be extracted.
Type and concentration of inflammatory cells present and selective biomarkers | The date of scheduled surgery assessed through the study completion, about two years
  The inflammatory profile of whole blood such as the quantity and type of circulating immune cells, e.g. complete blood count (CBC) with differential will be assessed using flow cytometry.A blood sample, about 10mL in volume, will be obtained at the preoperative waiting area immediately after IV placement.

SECONDARY OUTCOMES:
Perceived pain using a visual pain scale | ~2 weeks before surgery; 24, 36, 48, and 72 hours post-surgery before discharge; ~2 weeks after discharge
  standard Wong-Baker FACES® Pain Rating Scale of 0-10, 0 being no pain, 10 being worst pain
Perceived pain using the McGill pain scale | ~2 weeks before surgery; 24 hours post-surgery before discharge; ~2 weeks after discharge
  The McGill Pain Questionnaire (MPQ) is composed of 78 words. Respondents choose those that best describe their experience of pain.The McGill pain scale descriptors fall into four groups: sensory, affective, evaluative, and miscellaneous. Scores are tabulated by summing values associated with each word; scores range from 0 (no pain) to 78 (severe pain).
Anesthesia and pain management method | Within 1 week of the surgical visit
  Anesthesia method will be abstracted from the electronic medical records.
Opioid burden | Within 1 week of the surgical visit
  The total amount of analgesics administered will be abstracted from the electronic medical records.
Post-operative recovery and complications | Within 1 week of the surgical visit
  Incision site healing status, infection, and any complications will be abstracted from the electronic medical records.
Perceived pain during postsurgical recovery using the remote pain survey. | 1, 2, 3, 4 week post-discharge
  Investigator-developed pain survey that describes the pain level, location, and how it affects quality of life. The survey contains a pain scale from 0 to 10 with 0 being no pain and 10 being worst pain. The survey also contains non-numerical measures describing the location and impact of the pain.

CONTACTS AND LOCATIONS:
Overall Officials: Ala Nozari, MD PhD, Principal Investigator — Boston Medical Center, Anesthesiology
Locations (1):
- Boston Medical Center/Boston University Medical Campus, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No